CLINICAL TRIAL: NCT06397794
Title: Mixed Methods Study on Navigating Pregnancy and Parenthood With Lyme Disease
Brief Title: Navigating Pregnancy and Parenthood With Lyme Disease
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Collaborators: Clinical Trials Network for Lyme and Other Tick-Borne Diseases (Unknown); Steven & Alexandra Cohen Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: 00000932
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Lyme Disease; Post Treatment Lyme Disease; Chronic Lyme Disease; Tick-Borne Infections; Tick-Borne Diseases; Pregnancy Complications; Parenting
MeSH Terms: conditions — Lyme Disease; Post-Lyme Disease Syndrome; Tick-Borne Diseases; Pregnancy Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gestational parents with Lyme disease: Participants in this study will be enrolled following a screening call to assess their eligibility. All participants must report that they were diagnosed with acute Lyme disease, PTLDS, and/or Chronic Lyme by a health care provider while they were pregnant OR PTLDS/CL prior to becoming pregnant with ongoing symptoms during pregnancy.
  After being consented for the study, participants will then complete a set of online questionnaires and participate in a qualitative interview with a member of the research team.
  Interventions: Other: Quantitative surveys and qualitative interview

INTERVENTIONS:
Other: Quantitative surveys and qualitative interview — All participants will complete online surveys on topics including demographic and socioeconomic information, medical history (parent and child), pregnancy history, and mental health and well-being. They will then participate in a qualitative interview about their pregnancy and parenting experiences as gestational parents with Lyme disease.

SUMMARY:
This is a mixed methods study exploring the experiences of pregnancy and parenting among participants with Lyme disease. Eligible participants will have been diagnosed with Lyme disease (LD), post-treatment Lyme disease syndrome (PTLDS), and/or chronic Lyme (CL) either during or before a prior pregnancy. Participants will complete quantitative surveys on topics such as their medical history, their child(ren)'s development, and demographic information. They will then participate in a qualitative interview where they will be asked about their experiences with pregnancy and with parenting their child(ren) in the context of their condition.

DETAILED DESCRIPTION:
Patients with chronic conditions may experience the perinatal period and the experience of parenting differently than their healthy peers. The purpose of this study is to understand the lived experiences of pregnancy and parenting among gestational parents with Lyme disease.

Participants may be included in this study if they report having received a diagnosis of Lyme disease (LD), post-treatment Lyme disease syndrome (PTLDS), or chronic Lyme (CL) and they have given birth to at least one liveborn child. The investigators hypothesize that patients with LD/PTLDS/CL will experience unique challenges related to pregnancy, experiences in medical care settings, and their child's development.

Enrolled participants will complete a brief set of online quantitative questionnaires on topics such as their demographic characteristics, family information, Lyme disease histories, and mental health. The investigators will report on these data to illustrate similarities and differences between participants in the study for potentially relevant factors (e.g., timing of Lyme diagnosis relative to pregnancy, symptoms, mental health concerns). The questionnaires will be followed by an in-depth qualitative interview in English with each participant to learn about their experiences related to pregnancy and parenting with LD/PTLDS/CL, including specific questions about navigating the health care system, information seeking behaviors, and their child's development.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age and reside in the United States or Canada
* Diagnosed with acute Lyme disease, PTLDS, and/or Chronic Lyme by a health care provider while they were pregnant OR PTLDS/CL prior to becoming pregnant with ongoing symptoms during pregnancy

Exclusion Criteria:

* Under 18 years of age
* Live outside of the United States or Canada
* Never been diagnosed with Lyme disease by a medical provider
* Never been pregnant
* Never given birth to a liveborn infant
* Previously participated in a qualitative study about their experience with Lyme disease
* Do not want to agree to having their interviews audio recorded

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll up to 30 participants in this study, all of whom have been pregnant in the past and given birth to at least one liveborn child. There is no limit to the number of children a participant has, age of child(ren), or duration of Lyme-related symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Understand the lived experiences of pregnancy and parenting among gestational parents with LD, PTLDS, and/or CL | 3/20/2024 - 3/1/2025
  Semi-structured qualitative interviews will be conducted with parents with LD, PTLDS, and/or CL to understand their lived experience. The interviewer will follow a structured interview guide about participants' Lyme disease history, pregnancy, parenting experience, relationships, and their priorities. The interviewer will ask open-ended questions to understand participants' context and allow participants to share what they feel is important to them.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | 3/20/2024 - 3/1/2025
  Participants will complete the Edinburgh Postnatal Depression Scale (EPDS) prior to their qualitative interviews. The EPDS is a 10-question standardized postnatal depression screener.
General Anxiety Disorder-7 (GAD-7) | 3/20/2024 - 3/1/2025
  Participants will complete the General Anxiety Disorder-7 (GAD-7) screener prior to their qualitative interviews. The GAD-7 is a 7-question standardized assessment that measures severity of anxiety symptoms.
Parenting Stress Index 4th Edition, Short Form (PSI-4 SF) | 3/20/2024 - 3/1/2025
  Participants will complete the Parenting Stress Index 4th Edition, Short Form (PSI-4 SF) prior to their qualitative interviews. The PSI-4 SF is a standardized assessment that measures child and parent characteristics and stress experienced by a parent.
36-Item Short Form Survey (SF-36) | 3/20/2024 - 3/1/2025
  Participants will complete the36-Item Short Form Survey (SF-36) prior to their qualitative interviews. The SF-36 is a standardized quality of life assessment.
World Health Organization Disability Assessment Schedule (WHODAS 2.0) | 3/20/2024 - 3/1/2025
  Participants will complete the WHO Disability Assessment Schedule (WHODAS 2.0) prior to their qualitative interviews. The WHODAS 2.0 is a 36-question standardized measure of health and disability.
Posttraumatic Diagnostic Scale (PDS-5) | 3/20/2024 - 3/1/2025
  Participants will complete a modified version of the Posttraumatic Diagnostic Scale (PDS-5) prior to their qualitative interviews. The PDS-5 is a 24-question standardized measure of posttraumatic stress symptomatology. Participants will answer questions specific to their experience with Lyme disease.
Positive Affect and Well-Being Scale | 3/20/2024 - 3/1/2025
  Participants will complete the Positive Affect and Well-Being Scale prior to their qualitative interviews. The Positive Affect and Well-Being Scale is a 9-item measure of participants' sense of well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah B. Mulkey, MD, PhD, Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Participant enrollment screener — https://cri-datacap.org/surveys/?s=Y443RE43E43XN9D8